CLINICAL TRIAL: NCT05943067
Title: A Multi-center Phase I/II Trial of Memory T Cell Donor Lymphocyte Infusions After Transplantation of CliniMACS® TCRα/β and CD19 Depleted Stem Cell Grafts From Haploidentical Donors for Hematopoietic Cell Transplantation
Brief Title: CD45RA Depleted DLI After TCRα/β Depleted Haploidentical HCT
Acronym: CD45RADLIHaplo
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD45RADLIHaplo
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Other): Donor lymphocytes from allogeneic donors depleted of CD45RA lymphocytes.
  Interventions: Biological: CD45RA depleted donor lymphocyte infusion (DLI)

INTERVENTIONS:
Biological: CD45RA depleted donor lymphocyte infusion (DLI) — CD45RA depleted donor lymphocyte infusion (DLI) after TCRα/β depleted haploidentical HCT

SUMMARY:
The purpose of this clinical trial is to examine safety and toxicity of CD45RA depleted donor lymphocyte infusion (DLI) after transplantation of TCRα/β/CD19 depleted peripheral blood stem cells.

DETAILED DESCRIPTION:
Patients will undergo routine reduced intensity conditioning regimen and intravenous infusion of T-cell receptor alpha/beta (TCRα/β)/CD19 depleted peripheral blood stem cells (not content of clinical trial).

If no graft-versus-host disease (GVHD) occurs, patients receive the trial-related memory T cell donor lymphocyte infusion (DLI) on Day 30 after transplantation.

In a dose finding part (phase I) escalating doses will be applied in cohorts of three (three plus three design) patients with a maximum of 18 patients for three dose levels (dose level 1-3). A fourth lower dose level (dose level 0) is started, if >=2 out of 6 patients with dose level 1 develop aGVHD III/IV. The maximum tolerated dose (MTD) will be used for the confirmatory part (phase II) of the study.

ELIGIBILITY:
Inclusion Criteria:

Adult and pediatric patients with hematological malignancies in complete remission (CR), partial remission (PR) or with stable disease

* Acute myeloid leukemia (AML):

  * Patients with high-risk AML in first complete remission (CR1)
  * Patients with relapsed or primary therapy-refractory AML
* Acute lymphoid leukemia (ALL):

  * Patients with high-risk ALL in CR1
  * Patients with relapsed or primary refractory ALL
* Hodgkin's disease: Patients with relapsed or primary refractory Hodgkin's disease
* Non-Hodgkin's lymphoma: Patients with relapsed or primary refractory Non- Hodgkin's lymphoma
* Myelodysplastic Syndrome (MDS)/ Myeloproliferative Syndrome (MPS):

  °Patients with refractory MDS/MPS
* Multiple myeloma (MM): Patients with relapsed or refractory multiple myeloma

Exclusion Criteria:

* Age >65 years or <8 weeks
* Patients with progressive disease prior hematopoietic cell transplantation (HCT)
* <3 months after preceding HCT
* Treatment with T-cell or Interleukin-2 (IL-2) targeted medication (e.g. alemtuzumab, basiliximab) within 60 days prior to study product infusion
* Treatment with prednisolone at >2 mg/kg/day (or equivalent dosing of alternative glucocorticosteroids) at time of study product infusion.
* Known allergy/hypersensitivity to any component of the study product
* Treatment with another investigational drug within one month before inclusion
* History of neurological impairment (active seizures, severe peripheral neuropathy, signs of leukoencephalopathy, active Central Nervous System (CNS) infection) Note: For patients with heavy pretreatment with irradiation or intrathecal chemotherapy pre-transplant CNS MRI and neurological consultation are mandatory.
* Fungal infections with radiological and clinical progression
* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher than 400 U/L
* Chronic active viral hepatitis
* Ejection fraction <40% or Shortening fraction <20% on echocardiography. Patients with > grade II hypertension by Common Toxicity Criteria (CTC)
* Creatinine clearance below threshold defined for stem cell transplantation according to local clinical standard
* Respiratory failure necessitating supplemental oxygen
* HIV infection
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not willing to use an effective method of birth control during study treatment and for at least 12 months thereafter Note: Women of childbearing potential must have a negative serum pregnancy test at study entry.
* Concurrent severe or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which by assessment of the treating physician could compromise participation in the study
* Patients with a history of psychiatric illness or a condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol or unable to give informed consent

Ages: 8 Weeks to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phase I, dose escalation | 100 days
  Safety and toxicity of CD45RA depleted DLI as defined by infusional toxicities and acute GVHD grad III-IV.
Phase II, extension phase | 100 days
  Acute graft-versus-host disease grade III-IV defined as GVHD occurring within 100 days after HCT

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Children's Hospital University Clinic Tuebingen, Tübingen
  - University Hospital Tuebingen, Department of Hematology, Oncology, Immunology and Rheumatology, Tübingen

IPD SHARING:
Plan to Share IPD: No